CLINICAL TRIAL: NCT00306709
Title: Take HEED (Healthy Eating and Exercise Decisions)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Pamala Murphy, MD, Kaiser Permanente
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OH-04PMurp-01
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Obesity
Keywords: obesity; behavior change; cultural adaptations; weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teaching (Experimental)
  Interventions: Behavioral: culturally adapted behavior change

INTERVENTIONS:
Behavioral: culturally adapted behavior change — Behavior change strategies which have been modified to include spirituality, AA cultural materials and examples woven into the lesson plans, and sustained peer support.

SUMMARY:
This is a randomized intervention that examines the effect of culturally adapted weight loss program in African American (AA) females age 40-65. Evidence suggests that AA women are more successful with weight loss programs that are culturally tailored (Karanja, et al, 2002). Take HEED is a combination of 2 interventions, Therapeutic Lifestyle Changes Diet (TLC) from ATP-III and the CHANGE exercise program, which have shown success independently in previous clinical trials with AAs.

DETAILED DESCRIPTION:
Project/study objective(s), This is a randomized intervention that examines the effect of culturally adapted weight loss program in African American (AA) females age 40-65. Evidence suggests that AA women are more successful with weight loss programs that are culturally tailored (Karanja, et al, 2002). Take HEED is a combination of 2 interventions, Therapeutic Lifestyle Changes Diet (TLC) from ATP-III and the CHANGE exercise program, which have shown success independently in previous clinical trials with AAs.

Methods, The 21 month program (6 months active intervention and 15 months maintenance) is provided by a Nurse matched with the study participants for race, age, and gender. Take HEED uses behavior change strategies (Prochaska et al 1992) which have been modified to include spirituality, AA cultural materials and examples woven into the lesson plans, and sustained peer support. The diet has been modified to include calorie reductions, increased fruit/ vegetable and calcium intake, incorporation of AA ethnic recipes. Exercise has been culturally adapted featuring line- dancing, brisk walking and includes socialization time for development of strong interpersonal bonds that will encourage exercise in the participants. The control group receives KP's usual care which is a combination of nutrition classes and web based learning.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than 30
* African American
* 40-46 years old

Exclusion Criteria:

- bariatric surgery within the previous 5 years

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2005-02; Primary Completion 2007-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Examine the effect of culturally adapted weight loss program in African American (AA) females age 40-65

CONTACTS AND LOCATIONS:
Overall Officials: Pamala J Murphy, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Pemanente, Cleveland, Ohio, United States